CLINICAL TRIAL: NCT07181629
Title: Effectiveness of a Dysphagia Management Education Program for Caregivers of Stroke Patients Receiving Home Care
Brief Title: Dysphagia Management for Caregivers of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hicran Yıldız, Prof.Dr., Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H.Yıldız1
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Stroke ( 3 Months After Onset); Dysphagia; Palliative Care; Caregiver
Keywords: Stroke, dysphagia, caregiver, malnutrition, quality of life, caregiver burden
MeSH Terms: conditions — Stroke; Deglutition Disorders; Malnutrition; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Dysphagia Management Education
  Interventions: Behavioral: Dysphagia Management Education
- Control (Other)
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — The Personal Information Form, Mini Nutritional Assessment-Short Form (MNA-SF), Zarit Caregiver Burden Scale, Short Form-36 (SF-36) Quality of Life Questionnaire, and the Dysphagia Management Knowledge Form for Stroke Patients administered to caregivers of stroke patients at each interview (at 0, 1, and 3 months).
  Arms: Control
Behavioral: Dysphagia Management Education — The Personal Information Form, Mini Nutritional Assessment-Short Form (MNA-SF), Zarit Caregiver Burden Scale, Short Form-36 (SF-36) Quality of Life Questionnaire, and the Dysphagia Management Knowledge Form for Stroke Patients administered to caregivers of stroke patients at each interview (at 0, 1, and 3 months). The intervention group received dysphagia management training after the questionnaires were administered at the first meeting.
  Arms: Intervention

SUMMARY:
This randomized controlled experimental study was conducted to evaluate the effects of dysphagia management training provided to caregivers of stroke patients receiving home care. The sample size was determined using power analysis (n=84). Data were collected using the Personal Information Form, Mini Nutritional Assessment-Short Form (MNA-SF), Zarit Caregiver Burden Scale, Short Form-36 (SF-36) Quality of Life Questionnaire, and the Dysphagia Management Knowledge Form for Stroke Patients. Questionnaires were administered to both groups at baseline, the 1st month, and the 3rd month. The first application was administered to the intervention group before the education session.

DETAILED DESCRIPTION:
The experimental randomized controlled trial was conducted to evaluate the effects of dysphagia management training provided to caregivers of stroke patients receiving home care.The sample size was determined using power analysis (n=84). Patients who met the inclusion criteria were assigned to the experimental (n=42) and control (n=42) groups using a simple randomization technique. Data were collected using the the Personal Information Form, Mini Nutritional Assessment-Short Form (MNA-SF), Zarit Caregiver Burden Scale, Short Form-36 (SF-36) Quality of Life Questionnaire, and the Dysphagia Management Knowledge Form for Stroke Patients. Questionnaires were administered to both groups at baseline, the 1st month, and the 3rd month. The first application was administered to the intervention group before the education session.In data evaluation, percentages, means, independent t-tests, Pearson chi-square tests, Yates chi-square tests, repeated measures variance analysis (ANOVA), Pearson correlation tests, and Bonferroni tests were used.

ELIGIBILITY:
Inclusion Criteria:

Caregivers:

The caregiver must be between 18 and 60 years old. The caregiver must be willing and able to participate in the study. The caregiver must have at least a primary school education. The caregiver must be primarily responsible for the patient's care. The caregiver's Mini Mental Test score must be 25 or more. The caregiver's Beck Depression Inventory score must be below 17. The caregiver's Caregiver's Readiness to Care Scale score must be 16 or more.

Patients:

The patient's National Institutes of Health (NIH) Stroke Scale score must be 20 or less.

The patient must be between 18 and 60 years old. The patient must be receiving home care services. The patient must have been diagnosed with a stroke at least six months ago. The patient must have a Barthel index score of 90 or below.

Exclusion Criteria:

Caregivers:

The caregiver has a physical disability or serious health problem that makes caregiving difficult.

The caregiver has a Mini Mental Test score below 25 points. The caregiver has a Beck Depression Inventory score of 17 or higher. The caregiver has a Caregiver Readiness Scale score of 16 or lower. The caregiver has communication difficulties. The caregiver has a depression or psychiatric diagnosis. The caregiver is receiving psychotherapy/psychological support. The caregiver is taking antidepressants and/or anxiolytics. The caregiver has sensory loss related to vision or hearing.

Patients:

The patient has a Barthel index score of 91 or higher. The patient is receiving parenteral nutrition. The patient is receiving immunosuppressive therapy/immunotherapy and/or chemotherapy.

The patient has been diagnosed with cancer, an endocrine system disease, or a gastrointestinal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Care burden level | 0th month (1st day), 1st month and 3rd month
  The Zarit Care Burden Scale consists of 22 statements. As the score increases, the care burden also increases, and the maximum score is 88. Scores are graded as follows: (0-20) little/no burden, (21-40) moderate burden, (41-60) severe burden, and (61-88) excessive burden.
Quality of Life level | 0th month (1st day), 1st month and 3rd month
  SF-36 Quality of Life Scale: The scale consists of 36 questions and eight subscales. Each subscale is scored separately from 0 to 100. Higher scores indicate better health.
Nutritional Assessment level | 0th month (1st day), 1st month and 3rd month
  The MNA form consists of six questions. The maximum total score is 14. Individuals with a score of 12 or higher are considered to have adequate nutritional status, those with a score between 8 and 11 are at risk for malnutrition, and those with a score of 7 or less are considered malnourished.
Dysphagia management knowledge level | 0th month (1st day), 1st month and 3rd month
  The Dysphagia Management Knowledge Form for Stroke Patients Form for Stroke Patients consists of 26 statements, each answered with a true (0 point) or false (1 point) score. Scale scores range from 0 to 26. Higher scores indicate higher knowledge levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Simav Assoc. Prof. Dr. İsmail Karakuyu State Hospital Home Health Services Unit, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided